CLINICAL TRIAL: NCT03594630
Title: Organ Preservation With Active Surveillance After Chemoradiation in Rectal Cancer (OPTION)
Brief Title: Active Surveillance and Chemotherapy Before Surgery in Treating Participants With Stage II-III Rectal Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0549; NCI-2018-01142 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0549 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-20; First posted 2018-07-20 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v8; Stage IIA Rectal Cancer AJCC v8; Stage IIB Rectal Cancer AJCC v8; Stage IIC Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Watchful Waiting; Observation; Proctectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (surgical resection) (Active Comparator): Participants who have achieved clinical complete response undergo standard surgical resection.
  Interventions: Other: Questionnaire Administration; Procedure: Resection of Rectum
- Group II (active surveillance) (Experimental): Participants who have achieved clinical complete response receive active surveillance and consolidated chemotherapy for up to 4 months in the absence of disease progression or unacceptable toxicity. Participants with incomplete response or regrowth of tumor, undergo surgical resection as in Group I.
  Interventions: Drug: Chemotherapy; Other: Patient Observation; Other: Questionnaire Administration; Procedure: Resection of Rectum

INTERVENTIONS:
Drug: Chemotherapy — Receive chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
  Arms: Group II (active surveillance)
Other: Patient Observation — Receive active surveillance
  Other Names: Active Surveillance; deferred therapy; expectant management; observation; Watchful Waiting
  Arms: Group II (active surveillance)
Other: Questionnaire Administration — Ancillary studies
Procedure: Resection of Rectum — Undergo surgical resection
  Other Names: Proctectomy

SUMMARY:
This pilot trial studies how well active surveillance and chemotherapy before surgery work in treating participants with stage II-III rectal cancer. Active surveillance involves monitoring participants for additional tumor growth after receiving cancer treatment. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether deferring surgery after active surveillance and chemotherapy will work better in treating participants with stage II-III rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To quantify the rates of organ preservation and tumor regrowth with non-operative management of locally advanced rectal cancer in patients achieving a clinical complete response (cCR).

SECONDARY OBJECTIVES:

I. To correlate clinical, radiographic, and pathologic findings after neoadjuvant therapy for rectal cancer.

II. To determine the impact of active surveillance with deferral of surgery on oncologic outcomes.

III. To assess decision quality for patients with rectal cancer facing multiple treatment options.

IV. To explore the impact of patient-provider communication on patient decisions for surgical versus nonsurgical treatment decision for rectal cancer.

V. To assess safety of deferral of surgery in distal rectal cancer patients with possibility of cohort expansion to more proximal locally advanced rectal cancer patients.

CORRELATIVE OBJECTIVES:

I. Obtain tissue to monitor treatment response and any future biomarker analyses

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP I: Participants who have achieved clinical complete response undergo standard surgical resection.

GROUP II: Participants who have achieved clinical complete response receive active surveillance and consolidated chemotherapy for up to 4 months in the absence of disease progression or unacceptable toxicity. Participants with incomplete response or regrowth of tumor, undergo surgical resection as in Group I.

After the completion of study treatment, participants in Group I are followed up at 6 and 12 months, and then once a year for up to 3 years. Participants in Group II are followed up every 3 months for 18 months, every 6 months for 2 years, and then every year for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of rectal adenocarcinoma
* Eligible for curative resection of rectal adenocarcinoma
* Rectal tumor location =< 12 cm from the anal verge as determined by endoscopy or magnetic resonance imaging (MRI) (if endoscopy report is not available or deemed inadequate my treating oncologist)
* Nodal involvement confined to the radiation field
* Radiologically measurable or clinically evaluable disease as defined in the protocol
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0, 1 or 2
* Clinical Stage: Stage II and III. N2 disease is to be estimated as four or more lymph nodes that are >= 10 mm. Clinical staging should be estimated based on the combination of the following assessments: physical exam by the primary surgeon including digital rectal exam (DRE), computed tomography (CT) or positron emission tomography (PET)/CT scan of the chest/abdomen/pelvis and a pelvic MRI. If a pelvic MRI is performed, it is acceptable to perform CT of the chest/abdomen, omitting CT imaging of the pelvis. PET/CT is optional.
* No known contraindication to standard (fluoropyrimidine-based) pelvic chemoradiation (e.g. dihydropyrimidine dehydrogenase [DPD] deficiency)
* Patient of child-bearing potential is willing to employ adequate contraception during treatment and after treatment, as directed by treating clinical team
* Willing to provide written informed consent
* Willing to return to enrolling medical site for all study assessments

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease (IBD)
* Diagnosis of MSI-H colorectal cancer at time of consent
* Recurrent rectal cancer
* Tumor is causing symptomatic bowel obstruction (patients who have diverting ostomy are eligible)
* Any prior pelvic radiation
* Other invasive malignancy undergoing active treatment. Patients receiving prior treatment that precludes standard chemoradiation or ability to receive consolidation/adjuvant chemotherapy will be excluded from survival analyses
* Patients unwilling or unable to undergo pelvic MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall organ preservation rate | At 12 months
  The study will estimate overall organ preservation rate at 12 months and the corresponding 95% confidence interval (95% CI). The exact confidence interval will be computed when observed number of events is limited. The 12-month organ preservation rate corresponds to the proportion of patients alive and not having surgery within 12 months. The study will use Kaplan-Meier methods to estimate probability of overall organ preservation at 12 months at 12 months for all patients and for deferral patients respectively.
Local tumor regrowth rate | At 12 months
  The study will estimate local tumor regrowth rate at 12 months and the corresponding 95% confidence interval (95% CI). The exact confidence interval will be computed when observed number of events is limited. The 12-month organ preservation rate corresponds to the proportion of patients alive and not having surgery within 12 months. The study will use Kaplan-Meier methods to estimate probability of local tumor regrowth at 12 months for all patients and for deferral patients respectively.
Time to surgery or death | Up to 12 months
  The study will use Kaplan-Meier methods to estimate probability for deferral patients respectively.

SECONDARY OUTCOMES:
Decision quality assessment determined by European Organization for Treatment and Research of Cancer Quality of Life Questionnaire (EORTC-QLQ30+CR29) | Up to 3 years
  The aspects of the patient's decision making process will be documented and studied to assess what criteria, including the impact of patient-provider communication, seem to be driving the patients' decision to delay surgery or not. The decision evaluation questions such as decision quality survey, satisfaction with decision and anticipated regret questionnaire will be documented and summarized. Descriptive statistics will be used to summarize continuous variables and frequency and percentage will be used to tabulate categorical variables. The study will summarize quality of life measures, toxicity, surgical success rates, clinical, radiographic and pathologic findings, and exploratory comparisons among patient cohorts will be done.
Overall survival (OS) | Up to 5 years
  Overall survival will be estimated using Kaplan-Meier method.
Regression-free survival (RFS) | Up to 5 years
  Regression-free survival will be estimated using Kaplan-Meier method.
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 5 years
Surgical success rates | Up to 5 years
Radiographic Findings | Up to 5 years
  MRI performed.
Pathologic Findings | Up to 5 years
  Blood and tissue collected at various time points.

CONTACTS AND LOCATIONS:
Overall Officials: George Chang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org